CLINICAL TRIAL: NCT02841046
Title: The Application of Goal-directed Therapy With the Combination of Stroke Volume Variation and Cardiac Index as the Primary Judgment in Non-severe Patients Underwent Gastrointestinal Tumor Surgery
Brief Title: The Effect of Goal-directed Therapy Guided by Stroke Volume Variation and Cardiac Index in Non-severe Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lin Yang, Attending Physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2014]No.60
Record Dates: First submitted 2016-07-08; First posted 2016-07-21 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Fluid Therapy
Keywords: stroke volume variation; cardiac index; non-severe patients; gastrointestinal surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group cardiac index (Other): the treatment scheme of goal-directed fluid therapy(GDFT) use cardiac index（CI） as the primary judgment in group cardiac index,Patients in group cardiac index received a therapy with the goal of CI was no less than 2.5L•min-1•m-2 .
  Interventions: Device: cardiac index
- group Stroke Volume Variation (Experimental): the treatment scheme of goal-directed fluid therapy(GDFT) use Stroke Volume Variation（SVV）and cardiac index（CI）as the primary judgment in group Stroke Volume Variation,Patients in group Stroke Volume Variation received a therapy with SVV was less than 12% and CI was no less than 2.5L•min-1•m-2 .
  Interventions: Device: Stroke Volume Variation

INTERVENTIONS:
Device: cardiac index — group cardiac index（CI） and group Stroke Volume Variation（SVV） are different treatment schemes of goal-directed fluid therapy guided by SVV and CI,group cardiac index with CI as the primary judgment.
  Arms: group cardiac index
Device: Stroke Volume Variation — group cardiac index（CI） and group Stroke Volume Variation（SVV） are different treatment schemes of goal-directed fluid therapy guided by SVV and CI,group Stroke Volume Variation with the combination of SVV and CI as the primary judgment.
  Arms: group Stroke Volume Variation

SUMMARY:
To evaluate the application of fluid-infusion therapy with the combination of stroke volume variation (SVV) and cardiac index (CI) as the primary judgment in non-severe patients underwent resection of gastrointestinal tumor. Fifty patients (ASA Ⅰ-Ⅱ, 26-55 years old, cardiac functional gradingⅠ) scheduled for gastrointestinal tumor surgery were divided into two groups randomly: group C with CI as the primary judgment and group S with the combination of SVV and CI as the primary judgment.

DETAILED DESCRIPTION:
To evaluate the application of fluid-infusion therapy with the combination of stroke volume variation (SVV) and cardiac index (CI) as the primary judgment in non-severe patients underwent resection of gastrointestinal tumor.

Methods: Fifty patients (ASA Ⅰ-Ⅱ, 18-55 years old, cardiac functional gradingⅠ) scheduled for gastrointestinal tumor surgery were divided into two groups randomly: group C with CI as the primary judgment and group S with the combination of SVV and CI as the primary judgment. Patients in group C received a therapy with the goal of CI was no less than 2.5L•min-1•m-2 while SVV was less than 12% and CI was no less than 2.5L•min-1•m-2 in group S. Indexes including MAP、HR、CVP、CI、SVV were recorded at the moment after anaesthetized (T1), when skin was incised (T2), when the intestina was anastomosed (T3) and after the abdomen was closed (T4). SaO2、ScvO2 and plasma lactic were determined at T1 and T4 and DO2,VO2 and ERO2 during the surgery were calculated .The volume of fluid, vasoactive drugs use, the incidence of adverse cardiovascular events, the convalescence of intestinal peristalsis, hospital stay and postoperative complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status of grade I-II
* Cardiac function classification by NYHA of grade I
* without high risk factors according to the revised Lee cardiac risk index:

  1. High-risk type of surgery
  2. Ischemic heart disease
  3. History of congestive heart failure
  4. History of cerebrovascular disease
  5. Insulin therapy for diabetes
  6. Preoperative serum creatinine > 2.0 mg/dl
* undergoing gastrointestinal tumor surgery

Exclusion Criteria:

* Patients under 18 years or above 55 years
* patients with severe aortic regurgitation
* patients with permanent cardiac arrhythmias
* patients with intra-aortic balloon pump
* patients with severe pulmonary disease
* patients with hepatic or renal dysfunction
* patients undergoing emergency surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu HaiHua, doctor, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes
It should be discuss.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Della Rocca G, Pompei L. Goal-directed therapy in anesthesia: any clinical impact or just a fashion? Minerva Anestesiol. 2011 May;77(5):545-53. Epub 2011 Mar 1. PMID 21540811
- [Result] Futier E, Constantin JM, Petit A, Chanques G, Kwiatkowski F, Flamein R, Slim K, Sapin V, Jaber S, Bazin JE. Conservative vs restrictive individualized goal-directed fluid replacement strategy in major abdominal surgery: A prospective randomized trial. Arch Surg. 2010 Dec;145(12):1193-200. doi: 10.1001/archsurg.2010.275. PMID 21173294
- [Result] Cannesson M. Arterial pressure variation and goal-directed fluid therapy. J Cardiothorac Vasc Anesth. 2010 Jun;24(3):487-97. doi: 10.1053/j.jvca.2009.10.008. No abstract available. PMID 20022261
- [Result] Mathews L, Singh RK. Cardiac output monitoring. Ann Card Anaesth. 2008 Jan-Jun;11(1):56-68. doi: 10.4103/0971-9784.38455. PMID 18182765
- [Result] Cannesson M, Attof Y, Rosamel P, Joseph P, Bastien O, Lehot JJ. Comparison of FloTrac cardiac output monitoring system in patients undergoing coronary artery bypass grafting with pulmonary artery cardiac output measurements. Eur J Anaesthesiol. 2007 Oct;24(10):832-9. doi: 10.1017/S0265021507001056. Epub 2007 Aug 1. PMID 17666154
- [Result] Hofer CK, Senn A, Weibel L, Zollinger A. Assessment of stroke volume variation for prediction of fluid responsiveness using the modified FloTrac and PiCCOplus system. Crit Care. 2008;12(3):R82. doi: 10.1186/cc6933. Epub 2008 Jun 20. PMID 18570641
- [Result] Mayer J, Boldt J, Beschmann R, Stephan A, Suttner S. Uncalibrated arterial pressure waveform analysis for less-invasive cardiac output determination in obese patients undergoing cardiac surgery. Br J Anaesth. 2009 Aug;103(2):185-90. doi: 10.1093/bja/aep133. Epub 2009 May 29. PMID 19482857 (Retraction: PMID 21685126 Reilly C. Br J Anaesth. 2011 Jul;107(1):116-7)
- [Result] Vasdev S, Chauhan S, Choudhury M, Hote MP, Malik M, Kiran U. Arterial pressure waveform derived cardiac output FloTrac/Vigileo system (third generation software): comparison of two monitoring sites with the thermodilution cardiac output. J Clin Monit Comput. 2012 Apr;26(2):115-20. doi: 10.1007/s10877-012-9341-5. Epub 2012 Feb 17. PMID 22350311
- [Result] Samra T, Arya VK. Comparison of cardiac output estimation by FloTrac/Vigileo TM and intermittent pulmonary artery thermodilution in patient with Takayasu arteritis. Ann Card Anaesth. 2011 May-Aug;14(2):163-4. doi: 10.4103/0971-9784.81579. No abstract available. PMID 21636945
- [Result] Berkenstadt H, Margalit N, Hadani M, Friedman Z, Segal E, Villa Y, Perel A. Stroke volume variation as a predictor of fluid responsiveness in patients undergoing brain surgery. Anesth Analg. 2001 Apr;92(4):984-9. doi: 10.1097/00000539-200104000-00034. PMID 11273937
- [Result] Michard F, Alaya S, Zarka V, Bahloul M, Richard C, Teboul JL. Global end-diastolic volume as an indicator of cardiac preload in patients with septic shock. Chest. 2003 Nov;124(5):1900-8. doi: 10.1378/chest.124.5.1900. PMID 14605066
- [Result] Mayer J, Boldt J, Mengistu AM, Rohm KD, Suttner S. Goal-directed intraoperative therapy based on autocalibrated arterial pressure waveform analysis reduces hospital stay in high-risk surgical patients: a randomized, controlled trial. Crit Care. 2010;14(1):R18. doi: 10.1186/cc8875. Epub 2010 Feb 15. PMID 20156348
- [Result] Lang K, Suttner S, Boldt J, Kumle B, Nagel D. Volume replacement with HES 130/0.4 may reduce the inflammatory response in patients undergoing major abdominal surgery. Can J Anaesth. 2003 Dec;50(10):1009-16. doi: 10.1007/BF03018364. PMID 14656778 (Retraction: PMID 21792706 Miller DR. Can J Anaesth. 2011 Sep;58(9):883, 883-4)
- [Result] Lequeux PY, Bouckaert Y, Sekkat H, Van der Linden P, Stefanidis C, Huynh CH, Bejjani G, Bredas P. Continuous mixed venous and central venous oxygen saturation in cardiac surgery with cardiopulmonary bypass. Eur J Anaesthesiol. 2010 Mar;27(3):295-9. doi: 10.1097/EJA.0b013e3283315ad0. PMID 19935073
- [Result] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Cardiac Index | Group Stroke Volume Variation
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Cardiac Index | Group Stroke Volume Variation | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (7.9) | 39.7 (8.3) | 40.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 15 | 17 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Needed for Anal Exsufflation After Surgery
Description: record the number of days needed for anal exsufflation in non-severe patients after gastrointestinal tumor surgery
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group Cardiac Index | Group Stroke Volume Variation
Number analyzed (Participants) | 25 | 25
days | 3.8 (1.1) | 2.7 (1.2)

2. Secondary Outcome: the Incidence of Adverse Cardiovascular Events
Description: including hypertension,hypotension,tachycardia,bradycardia
Time Frame: during the surgery
Reporting Status: Not Posted

3. Secondary Outcome: Oxygen Delivery（DO2）
Description: oxygen delivery（DO2) in ml•min-1•m-2.Record the data of DO2 at the moment after anaesthetized immediately and at the moment when abdomen was closed.
Time Frame: during the surgery
Reporting Status: Not Posted

4. Secondary Outcome: Oxygen Consumption（VO2）
Description: oxygen delivery（VO2) in ml•min-1•m-2.Record the data of VO2 at the moment after anaesthetized immediately and at the moment when abdomen was closed.
Time Frame: during the surgery
Reporting Status: Not Posted

5. Secondary Outcome: Oxygen Extraction Rate（ERO2）
Description: oxygen extraction rate(ERO2) in percentage.Record the data of ERO2 at the moment after anaesthetized immediately and at the moment when abdomen was closed.
Time Frame: during the surgery
Reporting Status: Not Posted

6. Secondary Outcome: Number of Days in Hospital
Description: The number of days from the admission to hospital until the discharge from hospital
Time Frame: up to 10 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: The Volume of Crystalloid Infusion
Description: Volume of crystalloid infusion in milliliter.
Time Frame: during the surgery
Reporting Status: Not Posted

8. Other Pre Specified Outcome: The Volume of Colloid Infusion
Description: Volume of colloid infusion in milliliter.
Time Frame: during the surgery
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Complication After Surgery
Description: From the end of surgery to the time of discharge from hospital.including ileus,abdominal infection,infection of incisional wound,pulmonary infection
Time Frame: up to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Group Cardiac Index | Group Stroke Volume Variation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/25 | 1/25
Other Adverse Events (participants affected / at risk) | 2/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group Cardiac Index (N=25) | Group Stroke Volume Variation (N=25)
abdominal infection (Gastrointestinal disorders) | 4 | 1
ileus (Gastrointestinal disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group Cardiac Index (N=25) | Group Stroke Volume Variation (N=25)
infection of incisional wound (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT02841046/Prot_SAP_ICF_000.pdf